CLINICAL TRIAL: NCT06813859
Title: Monitored Effects of Physical Activity on Fetal Heart Rate by Using a Wireless Non-invasive Device
Status: Not yet recruiting | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01380
Record Dates: First submitted 2024-08-09; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exercise testing — incremental cycling test on a bicycle ergometer

SUMMARY:
Effect of acute exercise testing in pregnant athletes on maternal and fetal heart rate, fetal/maternal bloodflow and cardiotocogramm assessment.

DETAILED DESCRIPTION:
The aim of the study is to evaluate in a preliminary step the validity of fetal heart rate measurement with the "Nemo Healthcare Monitoring System" - a wireless non-invasive CTG device. Furthermore, we will determine the reliability for CTG measurements (intraobserver and interobserver reliability) and for ultrasound (intraobserver reliability). The device is approved for use on pregnant women and is regularly used as a CTG device for monitoring fetal heart rate and contractions during childbirth. If in the preliminary step the heart rate measurements with the "Nemo Fetal Monitoring System" provide valid and fetal heart rate results compared to the standard Doppler ultrasound method and provide a reliable detection of fetal heart rate deceleration the effects of phys-ical activity on fetal heart rate pattern and changes in fetal blood flow, placento-fetal and materno-placental blood supply rate will be investigated in the main part of the study in a larger study population.

It is hypothesized that CTG provides technically a valid and reliable continuous re-cording of fetal heart rate values, since fetal heart rate measurement under physical exertion has previously only been possible by intermittent but not continuous Dop-pler ultrasound. Furthermore, we will evaluate alterations in fetal heart rate pattern and changes in fetal blood flow, placento-fetal and materno-placental blood supply according to the level of exertion.

ELIGIBILITY:
Inclusion Criteria:

* Presence of signed informed consent form
* healthy pregnant active female over the age of 18 years and below 45 years
* sporting activity >4h/week on 2 or more weekdays
* single pregnancy, between 28+0 and 34+0 weeks of pregnancy

Exclusion Criteria:

* No signed informed consent form or revocation of consent
* pre-existing pregnancy complications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: pregnant athletes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
fetal heart rate | through exercise testing, an average of 90 minutes
  The fetal heart rate is continuously monitored via the CTG device during the entire performance test.

SECONDARY OUTCOMES:
Umbilical cord artery pulsatility index | through exercise testing, an average of 90 minutes
  (systolic velocity - diastolic velocity) / mean velocity
Umbilical cord artery resistance index | through exercise testing, an average of 90 minutes
  (systolic velocity - diastolic velocity) / systolic velocity
umbilical cord artery S/D ratio | through exercise testing, an average of 90 minutes
  (S = maximum systolic flow velocity; D = maximum diastolic flow velocity)
Medial cerebral artery pulsatility index | through exercise testing, an average of 90 minutes
  (systolic velocity - diastolic velocity) / mean velocity
Medial cerebral artery resistance index | through exercise testing, an average of 90 minutes
  (systolic velocity - diastolic velocity) / systolic velocity
medial cerebral artery peak systolic velocity | through exercise testing, an average of 90 minutes
  in cm/s
right and left uterine artery pulsatility index | through exercise testing, an average of 90 minutes
  (systolic velocity - diastolic velocity) / mean velocity
right and left uterine artery resistance index | through exercise testing, an average of 90 minutes
  (systolic velocity - diastolic velocity) / systolic velocity
cerebro-placental ratio | through exercise testing, an average of 90 minutes
  pulsatility index of the middle cerebral artery / pulsatility index of the umbilical artery
pregnancy complications | during pregnancy and up to12 weeks after birth
  incidence of pregnancy complications (yes/no);
birth complications | On the day the child is born
  incidence of birth complications (yes/no);
mode of delivery | On the day the child is born
  spontaneous birth vs. vacuum-assisted birth vs. forceps-assisted birth vs planned cesarean section vs. unplanned cesarean section
APGAR score | On the day the child is born
  APGAR score (1-10)
gestational age at birth | On the day the child is born
  gestational age at birth (in weeks and days);
pH value of the umbilical cord artery | On the day the child is born
  pH value of the umbilical cord artery mesured directly after birth
fetal admission to Neonatal Intensive Care Unit | up to 12 weeks
  admission (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Scherr, Prof. Dr. med., Study Chair — University Centre for Prevention and Sports Medicine, Department of Orthopaedics, Balgrist University Hospital, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No